CLINICAL TRIAL: NCT04239599
Title: Randomized Trial of Concomitant Hypofractionated IMRT Boost Versus Conventional Fractionated IMRT Boost for Localized High Risk Prostate Cancer
Brief Title: Trial of Hypofractionated IMRT Boost Versus Conventional IMRT Boost for Localized High Risk Prostate Cancer
Acronym: RCT-PHART2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCT- PHART2
Record Dates: First submitted 2019-10-29; First posted 2020-01-27 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — luprolide acetate gel depot; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Masking Description: This is a randomized Radiation trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypofractionation (Experimental): Hypofractionation: Using a one phase IMRT plan, the pelvic lymph nodes will be treated to a dose of 48 Gy in 25 fractions, while the prostate will be treated to a dose of 68 Gy in 25 fractions concomitantly (simulataneous integrated boost) + 18-36 months of Eligard Hormone injection.
  Interventions: Radiation: Hypofractionated IMRT Radiation treatment
- Standard Fractination (Active Comparator): Using 2 sequential IMRT plans, the pelvic lymph nodes and prostate will initially be treated to 46 Gy in 23 fractions, followed by a subsequent boost to the prostate to a total dose of 78 Gy + 18-36 months of Eligard Hormone injection.
  Interventions: Radiation: Hypofractionated IMRT Radiation treatment

INTERVENTIONS:
Radiation: Hypofractionated IMRT Radiation treatment
  Other Names: Eligard 22.5 mg (28.2 mg leuprolide acetate per syringe) [3-Month] for 18-36 months

SUMMARY:
Hypofractionation: 48 Gy in 25 fractions to pelvic lymph nodes while the prostate receives 68 Gy in 25 fractions concomitantly.

Standard Fractionation: pelvic lymph nodes and prostate will initially be treated to 46 Gy in 23 fractions, followed by a subsequent boost to the prostate to a total dose of 78 Gy over 39 fractions.

DETAILED DESCRIPTION:
Half the participants will receive using a one phase IMRT plan, the pelvic lymph nodes will be treated to a dose of 48 Gy in 25 fractions, while the prostate will be treated to a dose of 68 Gy in 25 fractions concomitantly (simulataneous integrated boost).

The other half of the participants will receive Standard fractionation using 2 sequential IMRT plans, the pelvic lymph nodes and prostate will initially be treated to 46 Gy in 23 fractions, followed by a subsequent boost to the prostate to a total dose of 78 Gy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained.
* Histologically confirmed diagnosis of adenocarcinoma of the prostate.
* Clinical stage T1-2 N0 M0, Gleason Score ≤ 7, PSA 20 - 100
* T1-2 N0 M0, Gleason Score 8 - 10, PSA ≤ 100
* T3 N0 M0, any Gleason Score, PSA ≤ 100

Exclusion Criteria:

* Patients with unilateral or bilateral hip replacement.
* Patients with active collagen vascular disease.
* Patients with active inflammatory bowel disease.
* Patients with previous radiotherapy to the pelvis.
* Patients with ataxia telangiectasia.
* Patients with nodal or distant metastases

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2011-03-31; Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 5 years
  The primary outcome for this study is PSA biochemical disease free survival at 5 years.

SECONDARY OUTCOMES:
Late GI and GU toxicities | 6 month post completion of treatment to end of 5 year follow up
  Number of participants with treatment-related adverse events as assessed by CTCAE v3.0, change from 6 months post treatment to end of 5 year follow-up.
Quality of life outcome: Expanded Prostate Index Composite (EPIC) | Baseline (start of treatment) to end of 5 year follow-up
  Measuring quality of life using the Expanded Prostate Cancer Index Composite (EPIC) questionnaire. The EPIC questionnaire consists of 50 questions. Each question is scored from 1-5, 5 being the better outcome and 1 being the worst outcome in most of the questions
Overall survival | Baseline to end of 5 year follow-up
  Overall survival comparing two treatment arms
Cancer specific survival | Baseline to end of 5 year follow-up
  Cancer specific survival comparing two treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Cheung, MD, Principal Investigator — Sunnybrook Health Sciences Centre

IPD SHARING:
Plan to Share IPD: No
There is no plan to share Individual Participant data. Results from the trial will be available through publications.